CLINICAL TRIAL: NCT03033953
Title: Effects of Native Whey and Milk Supplementation on Changes in Muscle Mass and Strength After 12 Weeks of Strength Training in Young and Elderly
Brief Title: Effects of Native Whey or Milk Supplementation on Adaptations to 12 Weeks of Strength Training in Young and Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian School of Sport Sciences (Other)
Collaborators: Tine (Industry); The Research Council of Norway (Other)
Responsible Party: Principal Investigator, Truls Raastad, Professor, Norwegian School of Sport Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: Tine 12wk
Record Dates: First submitted 2017-01-19; First posted 2017-01-27 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Healthy; Young; Elderly
MeSH Terms: interventions — Milk; Resistance Training

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Milk supplementation (Placebo Comparator): 11 (elderly) or 12 (young) weeks of strength training and daily supplementation of 2x20g milk protein.
  Interventions: Dietary Supplement: Milk; Other: Strength training
- Native whey (Experimental): 11 (elderly) or 12 (young) weeks of strength training and daily supplementation of 2x20g native whey protein.
  Interventions: Dietary Supplement: Native whey; Other: Strength training

INTERVENTIONS:
Dietary Supplement: Native whey
  Arms: Native whey
Dietary Supplement: Milk
  Arms: Milk supplementation
Other: Strength training

SUMMARY:
The aim of this study is to investigate the long term adaptations to 11 (elderly) or 12 (young) weeks of strength training when supplemented with native whey or milk. The investigators hypothesize that native whey will give greater increases in muscle hypertrophy and strength than milk.

DETAILED DESCRIPTION:
Increasing or maintaining muscle mass is of great importance for populations ranging from athletes to patients and elderly. Resistance exercise and protein ingestion are two of the most potent stimulators of muscle protein synthesis. Both the physical characteristic of proteins (e.g. different digestion rates of whey and casein) and the amino acid composition, affects the potential of a certain protein to stimulate muscle protein synthesis. Given its superior ability to rapidly increase blood leucine concentrations to high levels, whey is often considered the most potent protein source to stimulate muscle protein synthesis. Native whey protein is produced by filtration of unprocessed milk. Consequently, native whey has different characteristics than milk. Of special interest is the higher amounts of the highly anabolic amino acid leucine in native whey.

The higher levels of leucine can be of great interest for elderly individuals as some studies in elderly has shown an anabolic resistance to the effects of protein feeding and strength training. By increasing levels of leucine one might overcome this anabolic resistance in the elderly.

The aim of this double-blinded, randomized, partial cross-over study is to compare the changes in muscle hypertrophy and strength after a 11 (elderly) or 12 (young) week training intervention with daily supplementation of either 2x20g of native whey or milk proteins in young and elderly individuals. In order to explain potential differences between supplements an acute study investigating acute responses in blood amino acid concentrations and intracellular signalling is planned, in a subgroup of participants, before and after the training intervention.

The investigators hypothesize that native whey will induce greater muscle hypertrophy and strength gains than milk.

ELIGIBILITY:
Inclusion Criteria:

* Healthy in the sense that they can conduct training and testing
* Able to understand Norwegian language written and oral
* Between 20 and 45, or above 70 years of age

Exclusion Criteria:

* Diseases or injuries contraindicating participation
* Use of dietary supplements (e.g. proteins, vitamins and creatine)
* Lactose intolerance
* Allergy to milk
* Allergy towards local anesthetics (xylocain)

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2014-08; Primary Completion 2015-06 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Lean mass | Before the training intervention
  Measured by whole body dual x-ray absorptiometry (DXA)
Lean mass | After 11-12 weeks of strength training
  Measured by whole body dual x-ray absorptiometry (DXA)

SECONDARY OUTCOMES:
Thigh muscle cross sectional area | Before the training intervention
  Measured by magnetic resonance imaging (MRI)
Thigh muscle cross sectional area | After 11-12 weeks of strength training
  Measured by magnetic resonance imaging (MRI)
Pectoralis muscle cross sectional area | Before the training intervention
  Measured by magnetic resonance imaging (MRI)
Pectoralis muscle cross sectional area | After 11-12 weeks of strength training
  Measured by magnetic resonance imaging (MRI)
Arm cross sectional area | Before the training intervention
  Measured by magnetic resonance imaging (MRI)
Arm cross sectional area | After 11-12 weeks of strength training
  Measured by magnetic resonance imaging (MRI)
Thickness of the lateral vasti | Before the training intervention
  Measured by ultrasound
Thickness of the lateral vasti | After 11-12 weeks of strength training
  Measured by ultrasound
1 repetition maximum in leg press | Before the training intervention
1 repetition maximum in leg press | After 11-12 weeks of strength training
1 repetition maximum in bench press | Before the training intervention
1 repetition maximum in bench press | After 11-12 weeks of strength training
Ratio of phosphorylated to total ribosomal protein S6 kinase beta-1(P70S6K) change from baseline | 30 min before and 2 hours after exercise and protein supplement intake, before the training intervention
  Biopsies from m. Vastus Lateralis was analyzed by western blot
Ratio of phosphorylated to total ribosomal protein S6 kinase beta-1(P70S6K) change from baseline | 30 min before and 2 hours after exercise and protein supplement intake, after 11-12 weeks of strength training
  Biopsies from m. Vastus Lateralis was analyzed by western blot
Phosphorylation of phosphorylated to total eukaryotic elongation factor 2 (eEF-2) change from baseline | 30 min before and 2 hours after exercise and protein supplement intake, before the training intervention
  Biopsies from m. Vastus Lateralis was analyzed by western blot
Phosphorylation of phosphorylated to total eukaryotic elongation factor 2 (eEF-2) change from baseline | 30 min before and 2 hours after exercise and protein supplement intake, after 11-12 weeks of strength training
  Biopsies from m. Vastus Lateralis was analyzed by western blot
Phosphorylation of phosphorylated to total eukaryotic translation initiation factor 4E-binding protein 1 (4EBP-1) change from baseline | 30 min before and 2 hours after exercise and protein supplement intake, before the training intervention
  Biopsies from m. Vastus Lateralis was analyzed by western blot
Phosphorylation of phosphorylated to total eukaryotic translation initiation factor 4E-binding protein 1 (4EBP-1) change from baseline | 30 min before and 2 hours after exercise and protein supplement intake, after 11-12 weeks of strength training
  Biopsies from m. Vastus Lateralis was analyzed by western blot
Plasma amino acid concentration | 60 min before and 45, 60, 75 and 120 min after exercise and protein supplement intake, before the training intervention
Plasma amino acid concentration | 60 min before and 45, 60, 75 and 120 min after exercise and protein supplement intake, after 11-12 weeks of strength training
Muscle force generating capacity change from baseline | 15 min before, 10 min, 2.5 hours and 24 hours after exercise and protein supplement intake, before the training intervention
  Measured as unilateral isometric knee extension force (Nm) with 90° in the hip and knee joints.
Muscle force generating capacity change from baseline | 15 min before, 10 min, 2.5 hours and 24 hours after exercise and protein supplement intake, after 11-12 weeks of strength training
  Measured as unilateral isometric knee extension force (Nm) with 90° in the hip and knee joints.
Serum glucose | 60 min before and 45, 60, 75 and 120 min after exercise and protein supplement intake, before the training intervention
Serum glucose | 60 min before and 45, 60, 75 and 120 min after exercise and protein supplement intake, after 11-12 weeks of strength training
Serum insulin | 60 min before and 45, 60, 75 and 120 min after exercise and protein supplement intake, before the training intervention
Serum insulin | 60 min before and 45, 60, 75 and 120 min after exercise and protein supplement intake, after 11-12 weeks of strength training
Serum urea | 60 min before and 45, 60, 75 and 120 min after exercise and protein supplement intake, before the training intervention
Serum urea | 60 min before and 45, 60, 75 and 120 min after exercise and protein supplement intake, after 11-12 weeks of strength training
Serum creatine kinase | 60 min before and 45, 60, 75 and 120 min after exercise and protein supplement intake, before the training intervention
Serum creatine kinase | 60 min before and 45, 60, 75 and 120 min after exercise and protein supplement intake, after 11-12 weeks of strength training
Tumor necrosis factor alfa messenger ribonucleic acid (mRNA) | 30 min before exercise and protein intake, before training intervention
Tumor necrosis factor alfa mRNA | 2 hours after exercise and protein intake, before training intervention
Tumor necrosis factor alfa mRNA | 30 min before exercise and protein intake, after 11-12 weeks of strength training
Tumor necrosis factor alfa mRNA | 2 hours after exercise and protein intake, after 11-12 weeks of strength training
Interleukin 6 mRNA | 30 min before exercise and protein intake, before training intervention
Interleukin 6 mRNA | 2 hours after exercise and protein intake, before training intervention
Interleukin 6 mRNA | 30 min before exercise and protein intake, after 11-12 weeks of strength training
Interleukin 6 mRNA | 2 hours after exercise and protein intake, after 11-12 weeks of strength training
Interleukin 8 mRNA | 30 min before exercise and protein intake, before training intervention
Interleukin 8 mRNA | 2 hours after exercise and protein intake, before training intervention
Interleukin 8 mRNA | 30 min before exercise and protein intake, after 11-12 weeks of strength training
Interleukin 8 mRNA | 2 hours after exercise and protein intake, after 11-12 weeks of strength training
Nuclear Receptor Subfamily 4 Group A Member 2 mRNA | 30 min before exercise and protein intake, before training intervention
Nuclear Receptor Subfamily 4 Group A Member 2 mRNA | 2 hours after exercise and protein intake, before training intervention
Nuclear Receptor Subfamily 4 Group A Member 2 mRNA | 30 min before exercise and protein intake, after 11-12 weeks of strength training
Nuclear Receptor Subfamily 4 Group A Member 2 mRNA | 2 hours after exercise and protein intake, after 11-12 weeks of strength training
Interleukin 1b mRNA | 30 min before exercise and protein intake, before training intervention
Interleukin 1b mRNA | 2 hours after exercise and protein intake, before training intervention
Interleukin 1b mRNA | 30 min before exercise and protein intake, after 11-12 weeks of strength training
Interleukin 1b mRNA | 2 hours after exercise and protein intake, after 11-12 weeks of strength training
Interleukin 1 Receptor Antagonist mRNA | 30 min before exercise and protein intake, before training intervention
Interleukin 1 Receptor Antagonist mRNA | 2 hours after exercise and protein intake, before training intervention
Interleukin 1 Receptor Antagonist mRNA | 30 min before exercise and protein intake, after 11-12 weeks of strength training
Interleukin 1 Receptor Antagonist mRNA | 2 hours after exercise and protein intake, after 11-12 weeks of strength training
C-C Motif Chemokine Ligand 2 mRNA | 30 min before exercise and protein intake, before training intervention
C-C Motif Chemokine Ligand 2 mRNA | 2 hours after exercise and protein intake, before training intervention
C-C Motif Chemokine Ligand 2 mRNA | 30 min before exercise and protein intake, after 11-12 weeks of strength training
C-C Motif Chemokine Ligand 2 mRNA | 2 hours after exercise and protein intake, after 11-12 weeks of strength training
Interleukin 4 mRNA | 30 min before exercise and protein intake, before training intervention
Interleukin 4 mRNA | 2 hours after exercise and protein intake, before training intervention
Interleukin 4 mRNA | 30 min before exercise and protein intake, after 11-12 weeks of strength training
Interleukin 4 mRNA | 2 hours after exercise and protein intake, after 11-12 weeks of strength training
Interleukin 10 mRNA | 30 min before exercise and protein intake, before training intervention
Interleukin 10 mRNA | 2 hours after exercise and protein intake, before training intervention
Interleukin 10 mRNA | 30 min before exercise and protein intake, after 11-12 weeks of strength training
Interleukin 10 mRNA | 2 hours after exercise and protein intake, after 11-12 weeks of strength training
C-X-C Motif Chemokine Ligand mRNA | 30 min before exercise and protein intake, before training intervention
C-X-C Motif Chemokine Ligand mRNA | 2 hours after exercise and protein intake, before training intervention
C-X-C Motif Chemokine Ligand mRNA | 30 min before exercise and protein intake, after 11-12 weeks of strength training
C-X-C Motif Chemokine Ligand mRNA | 2 hours after exercise and protein intake, after 11-12 weeks of strength training
Cholesterol 25-Hydroxylase mRNA | 30 min before exercise and protein intake, before training intervention
Cholesterol 25-Hydroxylase mRNA | 2 hours after exercise and protein intake, before training intervention
Cholesterol 25-Hydroxylase mRNA | 30 min before exercise and protein intake, after 11-12 weeks of strength training
Cholesterol 25-Hydroxylase mRNA | 2 hours after exercise and protein intake, after 11-12 weeks of strength training
C-C Motif Chemokine Ligand 8 mRNA | 30 min before exercise and protein intake, before training intervention
C-C Motif Chemokine Ligand 8 mRNA | 2 hours after exercise and protein intake, before training intervention
C-C Motif Chemokine Ligand 8 mRNA | 30 min before exercise and protein intake, after 11-12 weeks of strength training
C-C Motif Chemokine Ligand 8 mRNA | 2 hours after exercise and protein intake, after 11-12 weeks of strength training
Interleukin 17D mRNA | 30 min before exercise and protein intake, before training intervention
Interleukin 17D mRNA | 2 hours after exercise and protein intake, before training intervention
Interleukin 17D mRNA | 30 min before exercise and protein intake, after 11-12 weeks of strength training
Interleukin 17D mRNA | 2 hours after exercise and protein intake, after 11-12 weeks of strength training
C-C Motif Chemokine Ligand 3 mRNA | 30 min before exercise and protein intake, before training intervention
C-C Motif Chemokine Ligand 3 mRNA | 2 hours after exercise and protein intake, before training intervention
C-C Motif Chemokine Ligand 3 mRNA | 30 min before exercise and protein intake, after 11-12 weeks of strength training
C-C Motif Chemokine Ligand 3 mRNA | 2 hours after exercise and protein intake, after 11-12 weeks of strength training
Peroxisome Proliferator-Activated Receptor Gamma, Coactivator 1 Alpha mRNA | 30 min before exercise and protein intake, before training intervention
Peroxisome Proliferator-Activated Receptor Gamma, Coactivator 1 Alpha mRNA | 2 hours after exercise and protein intake, before training intervention
Peroxisome Proliferator-Activated Receptor Gamma, Coactivator 1 Alpha mRNA | 30 min before exercise and protein intake, after 11-12 weeks of strength training
Peroxisome Proliferator-Activated Receptor Gamma, Coactivator 1 Alpha mRNA | 2 hours after exercise and protein intake, after 11-12 weeks of strength training
C-X-C Motif Chemokine Ligand 16 mRNA | 30 min before exercise and protein intake, before training intervention
C-X-C Motif Chemokine Ligand 16 mRNA | 2 hours after exercise and protein intake, before training intervention
C-X-C Motif Chemokine Ligand 16 mRNA | 30 min before exercise and protein intake, after 11-12 weeks of strength training
C-X-C Motif Chemokine Ligand 16 mRNA | 2 hours after exercise and protein intake, after 11-12 weeks of strength training
C-C Motif Chemokine Ligand 5 mRNA | 30 min before exercise and protein intake, before training intervention
C-C Motif Chemokine Ligand 5 mRNA | 2 hours after exercise and protein intake, before training intervention
C-C Motif Chemokine Ligand 5 mRNA | 30 min before exercise and protein intake, after 11-12 weeks of strength training
C-C Motif Chemokine Ligand 5 mRNA | 2 hours after exercise and protein intake, after 11-12 weeks of strength training
Nuclear Receptor Subfamily 4 Group A Member 3 mRNA | 30 min before exercise and protein intake, before training intervention
Nuclear Receptor Subfamily 4 Group A Member 3 mRNA | 2 hours after exercise and protein intake, before training intervention
Nuclear Receptor Subfamily 4 Group A Member 3 mRNA | 30 min before exercise and protein intake, after 11-12 weeks of strength training
Nuclear Receptor Subfamily 4 Group A Member 3 mRNA | 2 hours after exercise and protein intake, after 11-12 weeks of strength training
Uncoupling Protein 1 mRNA | 30 min before exercise and protein intake, before training intervention
Uncoupling Protein 1 mRNA | 2 hours after exercise and protein intake, before training intervention
Uncoupling Protein 1 mRNA | 30 min before exercise and protein intake, after 11-12 weeks of strength training
Uncoupling Protein 1 mRNA | 2 hours after exercise and protein intake, after 11-12 weeks of strength training
Matrix Metallopeptidase 9 mRNA | 30 min before exercise and protein intake, before training intervention
Matrix Metallopeptidase 9 mRNA | 2 hours after exercise and protein intake, before training intervention
Matrix Metallopeptidase 9 mRNA | 30 min before exercise and protein intake, after 11-12 weeks of strength training
Matrix Metallopeptidase 9 mRNA | 2 hours after exercise and protein intake, after 11-12 weeks of strength training
ATP Binding Cassette Subfamily A Member 1 mRNA | 30 min before exercise and protein intake, before training intervention
ATP Binding Cassette Subfamily A Member 1 mRNA | 2 hours after exercise and protein intake, before training intervention
ATP Binding Cassette Subfamily A Member 1 mRNA | 30 min before exercise and protein intake, after 11-12 weeks of strength training
ATP Binding Cassette Subfamily A Member 1 mRNA | 2 hours after exercise and protein intake, after 11-12 weeks of strength training
Leukocyte Differentiation Antigen CD36 mRNA | 30 min before exercise and protein intake, before training intervention
Leukocyte Differentiation Antigen CD36 mRNA | 2 hours after exercise and protein intake, before training intervention
Leukocyte Differentiation Antigen CD36 mRNA | 30 min before exercise and protein intake, after 11-12 weeks of strength training
Leukocyte Differentiation Antigen CD36 mRNA | 2 hours after exercise and protein intake, after 11-12 weeks of strength training
Toll Like Receptor 2 mRNA | 30 min before exercise and protein intake, before training intervention
Toll Like Receptor 2 mRNA | 2 hours after exercise and protein intake, before training intervention
Toll Like Receptor 2 mRNA | 30 min before exercise and protein intake, after 11-12 weeks of strength training
Toll Like Receptor 2 mRNA | 2 hours after exercise and protein intake, after 11-12 weeks of strength training
Nuclear Receptor Subfamily 1 Group H Member 3 mRNA | 30 min before exercise and protein intake, before training intervention
Nuclear Receptor Subfamily 1 Group H Member 3 mRNA | 2 hours after exercise and protein intake, before training intervention
Nuclear Receptor Subfamily 1 Group H Member 3 mRNA | 30 min before exercise and protein intake, after 11-12 weeks of strength training
Nuclear Receptor Subfamily 1 Group H Member 3 mRNA | 2 hours after exercise and protein intake, after 11-12 weeks of strength training
Solute Carrier Family 3 Member 2 mRNA | 30 min before exercise and protein intake, before training intervention
Solute Carrier Family 3 Member 2 mRNA | 2 hours after exercise and protein intake, before training intervention
Solute Carrier Family 3 Member 2 mRNA | 30 min before exercise and protein intake, after 11-12 weeks of strength training
Solute Carrier Family 3 Member 2 mRNA | 2 hours after exercise and protein intake, after 11-12 weeks of strength training
Solute Carrier Family 7 Member 5 mRNA | 30 min before exercise and protein intake, before training intervention
Solute Carrier Family 7 Member 5 mRNA | 2 hours after exercise and protein intake, before training intervention
Solute Carrier Family 7 Member 5 mRNA | 30 min before exercise and protein intake, after 11-12 weeks of strength training
Solute Carrier Family 7 Member 5 mRNA | 2 hours after exercise and protein intake, after 11-12 weeks of strength training
Solute Carrier Family 36 Member 1 mRNA | 30 min before exercise and protein intake, before training intervention
Solute Carrier Family 36 Member 1 mRNA | 2 hours after exercise and protein intake, before training intervention
Solute Carrier Family 36 Member 1 mRNA | 30 min before exercise and protein intake, after 11-12 weeks of strength training
Solute Carrier Family 36 Member 1 mRNA | 2 hours after exercise and protein intake, after 11-12 weeks of strength training
Solute Carrier Family 38 Member 2 mRNA | 30 min before exercise and protein intake, before training intervention
Solute Carrier Family 38 Member 2 mRNA | 2 hours after exercise and protein intake, before training intervention
Solute Carrier Family 38 Member 2 mRNA | 30 min before exercise and protein intake, after 11-12 weeks of strength training
Solute Carrier Family 38 Member 2 mRNA | 2 hours after exercise and protein intake, after 11-12 weeks of strength training
Muscle-Specific RING Finger Protein 1 mRNA | 30 min before exercise and protein intake, before training intervention
Muscle-Specific RING Finger Protein 1 mRNA | 2 hours after exercise and protein intake, before training intervention
Muscle-Specific RING Finger Protein 1 mRNA | 30 min before exercise and protein intake, after 11-12 weeks of strength training
Muscle-Specific RING Finger Protein 1 mRNA | 2 hours after exercise and protein intake, after 11-12 weeks of strength training
Atrogin-1 mRNA | 30 min before exercise and protein intake, before training intervention
Atrogin-1 mRNA | 2 hours after exercise and protein intake, before training intervention
Atrogin-1 mRNA | 30 min before exercise and protein intake, after 11-12 weeks of strength training
Atrogin-1 mRNA | 2 hours after exercise and protein intake, after 11-12 weeks of strength training
Forkhead Box Protein O1A mRNA | 30 min before exercise and protein intake, before training intervention
Forkhead Box Protein O1A mRNA | 2 hours after exercise and protein intake, before training intervention
Forkhead Box Protein O1A mRNA | 30 min before exercise and protein intake, after 11-12 weeks of strength training
Forkhead Box Protein O1A mRNA | 2 hours after exercise and protein intake, after 11-12 weeks of strength training
Forkhead Box O3 mRNA | 30 min before exercise and protein intake, before training intervention
Forkhead Box O3 mRNA | 2 hours after exercise and protein intake, before training intervention
Forkhead Box O3 mRNA | 30 min before exercise and protein intake, after 11-12 weeks of strength training
Forkhead Box O3 mRNA | 2 hours after exercise and protein intake, after 11-12 weeks of strength training
Myosin Heavy Chain 7 mRNA | 30 min before exercise and protein intake, before training intervention
Myosin Heavy Chain 7 mRNA | 2 hours after exercise and protein intake, before training intervention
Myosin Heavy Chain 7 mRNA | 30 min before exercise and protein intake, after 11-12 weeks of strength training
Myosin Heavy Chain 7 mRNA | 2 hours after exercise and protein intake, after 11-12 weeks of strength training
Myosin Heavy Chain 2 mRNA | 30 min before exercise and protein intake, before training intervention
Myosin Heavy Chain 2 mRNA | 2 hours after exercise and protein intake, before training intervention
Myosin Heavy Chain 2 mRNA | 30 min before exercise and protein intake, after 11-12 weeks of strength training
Myosin Heavy Chain 2 mRNA | 2 hours after exercise and protein intake, after 11-12 weeks of strength training
Myosin Heavy Chain 1 mRNA Myosin Heavy Chain 1 mRNA | 30 min before exercise and protein intake, before training intervention
Myosin Heavy Chain 1 mRNA Myosin Heavy Chain 1 mRNA | 2 hours after exercise and protein intake, before training intervention
Myosin Heavy Chain 1mRNA Myosin Heavy Chain 1 mRNA | 30 min before exercise and protein intake, after 11-12 weeks of strength training
Myosin Heavy Chain 1 mRNA Myosin Heavy Chain 1 mRNA | 2 hours after exercise and protein intake, after 11-12 weeks of strength training
Insulin Like Growth Factor 1 mRNA Myosin Heavy Chain 1 mRNA | 30 min before exercise and protein intake, before training intervention
Insulin Like Growth Factor 1 mRNA Myosin Heavy Chain 1 mRNA | 2 hours after exercise and protein intake, before training intervention
Insulin Like Growth Factor 1 mRNA Myosin Heavy Chain 1 mRNA | 30 min before exercise and protein intake, after 11-12 weeks of strength training
Insulin Like Growth Factor 1 mRNA Myosin Heavy Chain 1 mRNA | 2 hours after exercise and protein intake, after 11-12 weeks of strength training
Mast Cell Growth Factor mRNA Myosin Heavy Chain 1 mRNA | 30 min before exercise and protein intake, before training intervention
Mast Cell Growth Factor mRNA Myosin Heavy Chain 1 mRNA | 2 hours after exercise and protein intake, before training intervention
Mast Cell Growth Factor mRNA Myosin Heavy Chain 1 mRNA | 30 min before exercise and protein intake, after 11-12 weeks of strength training
Mast Cell Growth Factor mRNA Myosin Heavy Chain 1 mRNA | 2 hours after exercise and protein intake, after 11-12 weeks of strength training
Hepatocyte Growth Factor mRNA Myosin Heavy Chain 1 mRNA | 30 min before exercise and protein intake, before training intervention
Hepatocyte Growth Factor mRNA Myosin Heavy Chain 1 mRNA | 2 hours after exercise and protein intake, before training intervention
Hepatocyte Growth Factor mRNA Myosin Heavy Chain 1 mRNA | 30 min before exercise and protein intake, after 11-12 weeks of strength training
Hepatocyte Growth Factor mRNA Myosin Heavy Chain 1 mRNA | 2 hours after exercise and protein intake, after 11-12 weeks of strength training
Myostatin mRNA Myosin Heavy Chain 1 mRNA | 30 min before exercise and protein intake, before training intervention
Myostatin mRNA Myosin Heavy Chain 1 mRNA | 2 hours after exercise and protein intake, before training intervention
Myostatin mRNA Myosin Heavy Chain 1 mRNA | 30 min before exercise and protein intake, after 11-12 weeks of strength training
Myostatin mRNA Myosin Heavy Chain 1 mRNA | 2 hours after exercise and protein intake, after 11-12 weeks of strength training
Striated Muscle Activator Of Rho-Dependent Signaling mRNA Myosin Heavy Chain 1 mRNA | 30 min before exercise and protein intake, before training intervention
Striated Muscle Activator Of Rho-Dependent Signaling mRNA Myosin Heavy Chain 1 mRNA | 2 hours after exercise and protein intake, before training intervention
Striated Muscle Activator Of Rho-Dependent Signaling mRNA Myosin Heavy Chain 1 mRNA | 30 min before exercise and protein intake, after 11-12 weeks of strength training
Striated Muscle Activator Of Rho-Dependent Signaling mRNA Myosin Heavy Chain 1 mRNA | 2 hours after exercise and protein intake, after 11-12 weeks of strength training
JunB Proto-Oncogene, AP-1 Transcription Factor Subunit mRNA Myosin Heavy Chain 1 mRNA | 30 min before exercise and protein intake, before training intervention
JunB Proto-Oncogene, AP-1 Transcription Factor Subunit mRNA Myosin Heavy Chain 1 mRNA | 2 hours after exercise and protein intake, before training intervention
JunB Proto-Oncogene, AP-1 Transcription Factor Subunit mRNA Myosin Heavy Chain 1 mRNA | 30 min before exercise and protein intake, after 11-12 weeks of strength training
JunB Proto-Oncogene, AP-1 Transcription Factor Subunit mRNA Myosin Heavy Chain 1 mRNA | 2 hours after exercise and protein intake, after 11-12 weeks of strength training
Actin, Alpha 1, Skeletal Muscle mRNA Myosin Heavy Chain 1 mRNA | 30 min before exercise and protein intake, before training intervention
Actin, Alpha 1, Skeletal Muscle mRNA Myosin Heavy Chain 1 mRNA | 2 hours after exercise and protein intake, before training intervention
Actin, Alpha 1, Skeletal Muscle mRNA Myosin Heavy Chain 1 mRNA | 30 min before exercise and protein intake, after 11-12 weeks of strength training
Actin, Alpha 1, Skeletal Muscle mRNA Myosin Heavy Chain 1 mRNA | 2 hours after exercise and protein intake, after 11-12 weeks of strength training
Colony Stimulating Factor 3 mRNA Myosin Heavy Chain 1 mRNA | 30 min before exercise and protein intake, before training intervention
Colony Stimulating Factor 3 mRNA Myosin Heavy Chain 1 mRNA | 2 hours after exercise and protein intake, before training intervention
Colony Stimulating Factor 3 mRNA Myosin Heavy Chain 1 mRNA | 30 min before exercise and protein intake, after 11-12 weeks of strength training
Colony Stimulating Factor 3 mRNA Myosin Heavy Chain 1 mRNA | 2 hours after exercise and protein intake, after 11-12 weeks of strength training
Prostaglandin-Endoperoxide Synthase 2 mRNA Myosin Heavy Chain 1 mRNA | 30 min before exercise and protein intake, before training intervention
Prostaglandin-Endoperoxide Synthase 2 mRNA Myosin Heavy Chain 1 mRNA | 2 hours after exercise and protein intake, before training intervention
Prostaglandin-Endoperoxide Synthase 2 mRNA Myosin Heavy Chain 1 mRNA | 30 min before exercise and protein intake, after 11-12 weeks of strength training
Prostaglandin-Endoperoxide Synthase 2 mRNA Myosin Heavy Chain 1 mRNA | 2 hours after exercise and protein intake, after 11-12 weeks of strength training
TATA-Box Binding Protein mRNA Myosin Heavy Chain 1 mRNA | 30 min before exercise and protein intake, before training intervention
TATA-Box Binding Protein mRNA Myosin Heavy Chain 1 mRNA | 2 hours after exercise and protein intake, before training intervention
TATA-Box Binding Protein mRNA Myosin Heavy Chain 1 mRNA | 30 min before exercise and protein intake, after 11-12 weeks of strength training
TATA-Box Binding Protein mRNA Myosin Heavy Chain 1 mRNA | 2 hours after exercise and protein intake, after 11-12 weeks of strength training
Filamin B mRNA Myosin Heavy Chain 1 mRNA | 30 min before exercise and protein intake, before training intervention
Filamin B mRNA Myosin Heavy Chain 1 mRNA | 2 hours after exercise and protein intake, before training intervention
Filamin B mRNA Myosin Heavy Chain 1 mRNA | 30 min before exercise and protein intake, after 11-12 weeks of strength training
Filamin B mRNA Myosin Heavy Chain 1 mRNA | 2 hours after exercise and protein intake, after 11-12 weeks of strength training
Beta-2-Microglobulin mRNA Myosin Heavy Chain 1 mRNA | 30 min before exercise and protein intake, before training intervention
Beta-2-Microglobulin mRNA Myosin Heavy Chain 1 mRNA | 2 hours after exercise and protein intake, before training intervention
Beta-2-Microglobulin mRNA Myosin Heavy Chain 1 mRNA | 30 min before exercise and protein intake, after 11-12 weeks of strength training
Beta-2-Microglobulin mRNA Myosin Heavy Chain 1 mRNA | 30 min after exercise and protein intake, after 11-12 weeks of strength training
Fasting cholesterol (only in elderly) | Before training intervention
Fasting cholesterol (only in elderly) | After 11-12 weeks of strength training
Fasting triglycerides (only in elderly) | Before training intervention
Fasting triglycerides (only in elderly) | After 11-12 weeks of strength training
Fasting LDL (only in elderly) | Before training intervention
Fasting LDL (only in elderly) | After 11-12 weeks of strength training
Fasting HDL (only in elderly) | Before training intervention
Fasting HDL (only in elderly) | After 11-12 weeks of strength training

CONTACTS AND LOCATIONS:
Locations (1):
- Norwegian School of Sport Sciences, Oslo, Oslo County, Norway

IPD SHARING:
Plan to Share IPD: Undecided